CLINICAL TRIAL: NCT00145704
Title: Treatment of Childhood Cancer Therapy-induced Osteopenia in Growth Hormone Deficient Adult Survivors: Does Bisphosphonate Treatment Improve Bone Mineral Density?
Brief Title: Study of Adults With Low Growth Hormone Who Survived Childhood Cancer Where Treatment Caused Low Bone Density
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to low enrollment, participants are no longer being examined or treated
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNY UMU IRB # 4689
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-03

CONDITIONS: Osteopenia
Keywords: osteopenia; growth hormone deficiency; pediatric malignancy
MeSH Terms: conditions — Bone Diseases, Metabolic; Dwarfism, Pituitary | interventions — Risedronic Acid; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth Hormone only (Active Comparator): No bisphosphonate therapy given, participants will take Vitamin D 400 IU daily for 18 months, as well as calcium carbonate 500 mg twice a day for 18 months.
  Interventions: Dietary Supplement: Vitamin D supplement; Dietary Supplement: Calcium
- Growth Hormone & Bisphosphonate Therapy (Experimental): Bisphosphonate Therapy-Risedronate 35 mg once a week for 18 months, Vitamin D 400 IU daily for 18 months and calcium carbonate 500 mg twice daily for 18 months
  Interventions: Drug: bisphosphonate therapy (risedronate); Dietary Supplement: Vitamin D supplement; Dietary Supplement: Calcium

INTERVENTIONS:
Drug: bisphosphonate therapy (risedronate) — Bisphosphonate therapy given to patients with growth hormone deficiency
  Arms: Growth Hormone & Bisphosphonate Therapy
Dietary Supplement: Vitamin D supplement — Vitamin D given to patients with growth hormone deficiency
  Other Names: Over the counter Vitamin D 400 IU.
Dietary Supplement: Calcium — calcium supplement given to patients with growth hormone deficiency

SUMMARY:
The purpose of this project is to evaluate the hypothesis that bisphosphonate treatment given to growth hormone deficient patients (regardless of current growth hormone replacement therapy status and without changing that status) significantly increases total body bone mineral density during an eighteen month period of treatment combined with calcium and Vitamin D when compared to calcium and Vitamin D treatment alone.

DETAILED DESCRIPTION:
Adult patients with Dexa scan (bone scan) z-scores < -1.0 (meaning low bone density) in at least one site will be selected for randomization. All patients who qualify for randomization will undergo baseline bloodwork for serum bone specific alkaline phosphatase (BSAP) and n-terminal telopeptides of collagen (NTX) levels. Recent bloodwork obtained as part of their ongoing long-term Pediatric Oncology and/or Endocrine clinic follow-up evaluation will be reviewed to exclude any baseline correctable confounding causes of osteopenia (low bone density). All women of childbearing potential will have a pregnancy test.

For those patients already on growth hormone replacement therapy, growth hormone will be administered as per standard of care, with standard dose ranges adjusted based upon IGF-1(Insulin like growth factor) monitoring. Those patients not currently receiving growth hormone replacement therapy will not be placed on therapy as a part of this study. Patients on and off growth hormone replacement therapy will be randomized in a block design to the two treatment arms to assure equal numbers in each treatment arm. The bisphosphonate to be utilized will be provided to the Arm II patients at no charge. All Arm II patients will receive the same bisphosphonate regimen, Risedronate 35 mg per oral once weekly for 18 months. All patients on arms I and II will also receive Vitamin D (400 IU p.o. daily) and calcium carbonate (500 mg p.o. twice daily) free of charge for eighteen months.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficiency as a complication of treatment for pediatric malignancy
* Dexa (bone densitometry)with z-scores of < -1.0 in at least one site

Exclusion Criteria:

* Dexa (bone densitometry)with z-scores < -1.0 in at least one site
* Subjects <18 years old
* Pregnant or lactating patients
* Any contraindication for or unwillingness to consider bisphosphonate treatment
* Inability or unwillingness to undergo bone density evaluation
* Other correctable causes of decreased bone mineral density

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2002-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult pts from Upstate Med Univ who have known growth hormone deficiency as a complication of treatment for pediatric malignancy will be selected after chart review from their Kids Not on Treatment(KNOT)Clinic records prior to their routine follow up appt.Pts will receive info about this study on their routine f/w up appts at the KNOT Clinic.
Groups:
- Bisphosphonate and Growth Hormone: bisphosphonate use and growth hormone use
- Growth Hormone Only: Growth hormone only, no bisphosphonate will be used
Period: Overall Study
Arm/Group | Bisphosphonate and Growth Hormone | Growth Hormone Only
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Bisphosphonate and Growth Hormone Use: bisphosphonate use and growth hormone use
- Growth Hormone Only: Growth hormone use only, no bisphosphonate used
- Total: Total of all reporting groups
Arm/Group | Bisphosphonate and Growth Hormone Use | Growth Hormone Only | Total
Number analyzed (Participants) | 3 | 3 | 6
Age Continuous [Median (Full Range); unit: years] | 25 [18 to 40] | 25 [18 to 40] | 25 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Bone Mineral Density During an 18 Month Period
Description: For those patients already on growth hormone replacement therapy, growth hormone will be administered as per standard of care, with standard dose ranges adjusted based upon IGF-1 monitoring. Those patients not currently receiving growth hormone replacement therapy will not be placed on therapy as a part of this study. Patients on and off growth hormone replacement therapy will be randomized in a block design to the two treatment arms to assure equal numbers in each treatment arm. The bisphosphonate to be utilized will be provided to the Arm II patients at no charge. All Arm II patients will receive the same bisphosphonate regimen, Risedronate 35 mg per oral once weekly for 18 months. All patients on arms I and II will also receive Vitamin D (400 IU p.o. daily) and calcium carbonate (500 mg p.o. twice daily) free of charge for eighteen months.
Time Frame: 18 months
Population: Data analyis halted, due to low enrollment,no outcomes to report
Arm/Group | Bisphosphonate and Growth Hormone Use | Growth Hormone Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: May, 2002 to October 2008
Arm/Group | Bisphosphonate and Growth Hormone Use | Growth Hormone Only
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment, and lost to follow up of three subjects. Data was limited and therefore not reviewed/analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No